CLINICAL TRIAL: NCT02098447
Title: Evaluation of Electrical Auricular Vagal Nerve Stimulation Effects on Parameters of Wound Healing in Chronic Diabetic Wounds - Pilot Study
Brief Title: Pilot Study on Auricular Vagus Nerve Stimulation Effects in Chronic Diabetic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Vienna University of Technology (Other)
Responsible Party: Principal Investigator, Dr. Jozsef Constantin Széles, Dr.med., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PS 01/2014
Record Dates: First submitted 2014-03-20; First posted 2014-03-28 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Chronic Diabetic Foot Ulcers
Keywords: vagus nerve stimulation effects on heart rate variability and peripheral blood perfusion

ARMS (1):
- auricular vagal nerve stimulation (Experimental): Study participants (healthy and diabetics) are treated with auricular vagal nerve stimulation using four needle electrodes connected to an electrical stimulation device (PrimeStim). After an acclimatization phase the stimulation is turned on for 20 minutes followed by 20 minutes of paused stimulation, 20 minutes of stimulation, and another 10 minutes paused stimulation. This intervention is repeated on four consecutive days. Needle electrodes stay fixed over the whole study period.
  Two different stimulation schemes are tested, each being assessed twice in random order. Stimulation amplitudes are adjusted with respect to a distinct but comfortable sensation at the auricle.
  During the described protocol various biosignals are continuously recorded, including ECG, respiration, blood perfusion, oxygen saturation, transcutaneous oxygen tension, blood pressure and skin temperature.
  Interventions: Device: PrimeStim

INTERVENTIONS:
Device: PrimeStim

SUMMARY:
The purpose of this pilot study is to evaluate the effect of auricular autonomous nervous system stimulation on vital parameters of wound healing in diabetics. It is investigated if auricular vagal nerve stimulation has an effect on heart rate variability as well as peripheral local blood perfusion, and if this effect depends on the health status of the study participants (diseased/healthy).

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus type 2
* ulcus cruris (plantar)
* min. 6 weeks of standard wound therapy without success
* intact big toe on wound side

Exclusion Criteria:

* participation in a clinical trial in the last 5 weeks
* confounding medical treatment, e.g. prostaglandin
* vascular diseases other than peripheral arterial occlusive disease
* diseases which may affect the autonomous nervous system or wound healing, except diabetic concomitant diseases (e.g., polyneuropathy, angiopathy)
* drug abuse
* active implanted devices
* pregnancy or nursing

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04-13 (Actual); Study Completion 2015-04-13 (Actual)

PRIMARY OUTCOMES:
change in heart rate variability (HRV) related to physiological state (diabetics/healthy) | within 4 days of intervention
  Heart rate variability will be assessed as, e.g., standard deviation in heart rate over a time window of 5 minutes (30 seconds overlap).
  Changes in mean value and standard deviation of heart rate variability between healthy and diabetic patients will be assessed using statistical tests.
change in local blood perfusion index (BPI) related to physiological state (diabetics/healthy) | within 4 days of intervention
  Blood perfusion index at the foot will be assessed as peak-peak amplitude (systolic to diastolic) divided by the mean signal value of optically measured blood perfusion.
  Changes in mean value and standard deviation of local blood perfusion index between healthy and diabetic patients will be assessed using statistical tests.

SECONDARY OUTCOMES:
Change in HRV and local BPI due to distinct stimulation patterns | within 4 days of intervention
  Two distinct stimulation patterns are tested during intervention.
  Changes in mean value and standard deviation of HRV/BPI due to these stimulation patterns will be assessed using statistical tests.
Change of local BPI in upper and lower extremities | within 4 days of intervention
  Local BPI is assessed using optical sensors on the foot and the finger of participants.
  Changes in mean value of BPI are analyzed using statistical tests.
Changes in blood pressure | within 4 days of intervention
  Blood pressure is continuously measured using inflatable finger cuffs.
Changes in respiratory activity | within 4 days of intervention
  Respiratory activity is monitored using a respiratory belt.
Changes in oxygen saturation of the toe and wound | within 4 days of intervention
Changes in partial transcutaneous oxygen pressure of the wound region | within 4 days of intervention
Changes in foot skin temperature | within 4 days of intervention
Changes of C reactive protein- and leukocyte-concentration in serum | within 4 days of intervention
Tolerance of stimulation | within 4 days of intervention
  Tolerance of stimulation is assessed by survey.
Perception of Stimulation | within 4 days of intervention
  Perception of stimulation is assessed by survey.
Adverse effects of stimulation | within 4 days of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jozsef C Széles, Dr.med., Principal Investigator — University Clinic for Surgery, Department of Transplantation, Medical University Vienna
Locations (1):
- University Clinic for Surgery, Department of Transplantation, Medical University Vienna, Vienna, Vienna, Austria